CLINICAL TRIAL: NCT06947915
Title: Co-producing a Novel Model an Outcome Framework for the Implementation of Falls Management in Care Home Settings.
Acronym: CHAFFINCH
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22011
Record Dates: First submitted 2025-04-04; First posted 2025-04-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Old Age; Long Term Care Facility; Fall Prevention
Keywords: long term care; falls management
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stakeholder: Stakeholder across the ICS: Key stakeholders within an ICS system including:
  carers, registered health professionals, managers and owners/executives from care homes commissioners, health care professionals and regulators involved in care home and falls management pathways residents living in care homes relatives of residents living in care homes
  Interventions: Other: Co-design workshop
- Care home staff: Any member of staff working in the case study care homes
  Interventions: Other: Survey; Other: Interview

INTERVENTIONS:
Other: Co-design workshop — Co-design workshops to develop the implementation model
  Groups: Stakeholder
Other: Survey — Survey of care staff knowledge and confidence
  Groups: Care home staff
Other: Interview — Interview to explore care staff experience of the falls management support
  Groups: Care home staff

SUMMARY:
AIM: To co-produce a novel model for implementation of falls management for older people living in care homes

SECONDARY OBJECTIVES

Component One Objectives:

Primary :To co-produce a novel model for the implementation of falls management in care homes Secondary

* To facilitate a series of co-production workshops with representation of key stakeholders
* To co-produce a novel implementation model for falls management
* To co-produce an outcomes framework to evaluate the implementation model
* To explore the feasibility of delivering the model and using the outcomes framework across Nottingham and Nottinghamshire Integrated Care Systems (ICSs)

Component Two Objectives:

* To evaluate how and the extent to which co-production occurs during the process of developing a novel model and an outcomes framework for the implementation for falls management in care homes
* To reflect on challenges and facilitators of using co-production approaches in this context
* To evaluate how care home residents can be supported to voice their priorities within the process.

DETAILED DESCRIPTION:
Component One: Co-production of the implementation model and outcomes framework A series of co-production workshops will be undertaken using a systemic action research methodology to develop and explore the feasibility of a novel implementation model and outcomes framework. This will involve three small workshop groups consisting of residents and relatives, care home staff only, and representatives from ICS partner organisations. All participants will be invited to attend a multi-stakeholder workshop in the later stages of the process to share ideas. Data collected for component one will be collected by the PI and PhD student. The novel model will be co-produced as part of this project but may include activities such as a care home audit programme, a reporting process, training and education and a community of practice. Following co-production of the model it will be delivered across Nottinghamshire ICB and refined in line with the systemic action research process.

Component Two: Evaluating the co-production process A process evaluation will be undertaken to explore how and the extent to which co-production occurs in component one, including reflection on challenges and facilitators, and how resident involvement is supported. Data collected for component two will be collected by the PhD student.

ELIGIBILITY:
Inclusion Criteria:

- Key stakeholders within an ICS system including: carers, registered health professionals, managers and owners/executives from care homes commissioners, health care professionals and regulators involved in care home and falls management pathways, residents living in care homes relatives of residents living in care homes

* 18 years and over (no upper age limit)
* Any member of staff working in the 10 case study care homes in Nottinghamshire

Exclusion Criteria:

* Unable to read and understand written English
* Lack of capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Care home staff, residents and ICS stakeholders
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Key features of the falls management implementation model and outcomes framework using thematic analysis from the co-design workshops through study completion anticipated at 18 months | From enrolment to the end of the co-design workshops at 12 months
  The data collected to address this primary includes:
  * The number of workshops, location, duration and range of stakeholders attending
  * Summary of key themes from each meeting drawn together from flipcharts, online flipchart programmes such as padlet and field notes
  * Cross-comparison of themes between the stakeholder groups
  * Record of between meeting activities to describe the types of information and activities undertaken
  * List of problems and potential solutions
  * Facilitator maintained notes on the decisions made in developing the model and the factors influencing the decisions
  * Description of the key features of the model Description of outcomes framework

CONTACTS AND LOCATIONS:
Overall Officials: Katie Robinson, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small number of participants

REFERENCES:
- [Result] Hallam-Bowles F, Kilby A, Gordon A, Timmons S, Logan P, Rees L, Lawry W; CHAFFINCH stakeholder group; Robinson K. A Qualitative Evaluation Exploring Co-Production of Falls Management in Care Homes. Health Expect. 2025 Dec;28(6):e70500. doi: 10.1111/hex.70500. PMID 41261769
- See also: Study webpage — https://www.nuh.nhs.uk/chaffinch-